CLINICAL TRIAL: NCT05124197
Title: Safety and Efficacy of a Strategy Extending Duration of Prone Position in COVID-19-related ARDS Patients. a Retrospective Monocentric Observational Study
Brief Title: Extended Prone Position Duration COVID-19-related ARDS: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care Medicine, Head ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR10
Record Dates: First submitted 2021-11-15; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Pressure Ulcer; Respiratory Distress Syndrome, Acute; Hypoxemic Respiratory Failure; COVID-19 Acute Respiratory Distress Syndrome
Keywords: prone position; mechanical ventilation
MeSH Terms: conditions — Pressure Ulcer; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of ICU patients with COVID-19 related ARDS requiring at least one extended PP session: patients with COVID-19 related ARDS requiring prone position because of profound hypoxemia were applied the investigators' strategy to extend duration of prone position: after being turned prone, they spent at least two complete nights in prone position before being turned to supine position
  Interventions: Other: prone position

INTERVENTIONS:
Other: prone position — extension of prone position duration

SUMMARY:
Prone position (PP) is standard of care for mechanically ventilated patients with severe acute respiratory distress syndrome in the intensive care unit (ICU). Recommendations suggest PP durations of at least 16 hours. In 2020, COVID-19 pandemic led to a great number of patients requiring mechanical ventilation and PP in the ICU. Risk of ICU staff viral contamination and work overload led to prolongation of PP duration up to 48 hours. Here investigators report outcomes of prolonged PP sessions in terms of skin complications (pression injuries) and ventilatory improvement.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a severe condition in which diffuse ventilation/perfusion mismatching and intra-pulmonary shunt are responsible for profound hypoxemia. In patients with severe ARDS, prone position (PP) improves oxygenation and reduces mortality. Recommendations suggest that PP sessions should last at least 16 consecutive hours. Safety concern is mainly related to the risk of pressure injuries.

In 2020, COVID-19 pandemic led to a great number of patients requiring mechanical ventilation (MV) and PP in the Intensive Care Units (ICUs) worldwide.

In the ICU of Louis Mourier hospital (Colombes, France) investigators decided upon a strategy whereby PP sessions duration was extended up to 48 hours in patients with COVID-19-related ARDS, so as to minimize the number and workload of turning procedures, limit staff exposure to viral contamination, and avoid turning patients during night shifts.

Here, investigators aim to report incidence of skin complications (pression injuries) in patients who underwent at least one prolonged PP session. Secondary objective was to evaluate evolution of ventilatory parameters with prolonged PP sessions.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 proven by PCR-testing of respiratory specimen
* Acute respiratory distress syndrome (Berlin definition) requiring invasive mechanical ventilation and prone position
* at least one session of prolonged prone position (that includes two consecutive nights in prone position)

Exclusion Criteria:

* transfer to another ICU facility after initial admission (inter-regional regulation of ICU beds' availability)

  * Incomplete or missing medical file
  * Refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult, ICU, COVID-19 related ARDS patients with profound hypoxemia requiring invasive mechanical ventilation and prone position
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of skin complications (pressure injuries) | from first prone position session to Day-28 or ICU discharge, whichever comes first
  overall and per stage (from stage 1 to stage 4) incidence of pressure injuries

SECONDARY OUTCOMES:
arterial blood gases | through each prone position session, that lasts an average of 39 hours: before session (T0), during session (T1) and immediately after session (T2)
  changes in arterial blood gases (partial pressure in oxygen, carbon dioxide and pH)
plateau pressure | through each prone position session, that lasts an average of 39 hours: before session (T0), during session (T1) and immediately after session (T2)
  teleinspiratory pause pressure
driving pressure | through each prone position session, that lasts an average of 39 hours: before session (T0), during session (T1) and immediately after session (T2)
  plateau minus positive end-expiratory pressure
respiratory compliance system | through each prone position session, that lasts an average of 39 hours: before session (T0), during session (T1) and immediately after session (T2)
  volume over pressure ratio of the respiratory system
positive end-expiratory pressure | through each prone position session, that lasts an average of 39 hours: before session (T0), during session (T1) and immediately after session (T2)
  positive end-expiratory pressure
inspired oxygen fraction | through each prone position session, that lasts an average of 39 hours: before session (T0), during session (T1) and immediately after session (T2)
  inspired oxygen fraction

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Assistance Publique - Hôpitaux de Paris, Colombes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Papazian L, Aubron C, Brochard L, Chiche JD, Combes A, Dreyfuss D, Forel JM, Guerin C, Jaber S, Mekontso-Dessap A, Mercat A, Richard JC, Roux D, Vieillard-Baron A, Faure H. Formal guidelines: management of acute respiratory distress syndrome. Ann Intensive Care. 2019 Jun 13;9(1):69. doi: 10.1186/s13613-019-0540-9. PMID 31197492
- [Background] Nasa P, Azoulay E, Khanna AK, Jain R, Gupta S, Javeri Y, Juneja D, Rangappa P, Sundararajan K, Alhazzani W, Antonelli M, Arabi YM, Bakker J, Brochard LJ, Deane AM, Du B, Einav S, Esteban A, Gajic O, Galvagno SM Jr, Guerin C, Jaber S, Khilnani GC, Koh Y, Lascarrou JB, Machado FR, Malbrain MLNG, Mancebo J, McCurdy MT, McGrath BA, Mehta S, Mekontso-Dessap A, Mer M, Nurok M, Park PK, Pelosi P, Peter JV, Phua J, Pilcher DV, Piquilloud L, Schellongowski P, Schultz MJ, Shankar-Hari M, Singh S, Sorbello M, Tiruvoipati R, Udy AA, Welte T, Myatra SN. Expert consensus statements for the management of COVID-19-related acute respiratory failure using a Delphi method. Crit Care. 2021 Mar 16;25(1):106. doi: 10.1186/s13054-021-03491-y. PMID 33726819
- [Background] Sud S, Friedrich JO, Adhikari NK, Taccone P, Mancebo J, Polli F, Latini R, Pesenti A, Curley MA, Fernandez R, Chan MC, Beuret P, Voggenreiter G, Sud M, Tognoni G, Gattinoni L, Guerin C. Effect of prone positioning during mechanical ventilation on mortality among patients with acute respiratory distress syndrome: a systematic review and meta-analysis. CMAJ. 2014 Jul 8;186(10):E381-90. doi: 10.1503/cmaj.140081. Epub 2014 May 26. PMID 24863923
- [Background] Labeau SO, Afonso E, Benbenishty J, Blackwood B, Boulanger C, Brett SJ, Calvino-Gunther S, Chaboyer W, Coyer F, Deschepper M, Francois G, Honore PM, Jankovic R, Khanna AK, Llaurado-Serra M, Lin F, Rose L, Rubulotta F, Saager L, Williams G, Blot SI; DecubICUs Study Team; European Society of Intensive Care Medicine (ESICM) Trials Group Collaborators. Prevalence, associated factors and outcomes of pressure injuries in adult intensive care unit patients: the DecubICUs study. Intensive Care Med. 2021 Feb;47(2):160-169. doi: 10.1007/s00134-020-06234-9. Epub 2020 Oct 9. PMID 33034686
- [Background] Gaudry S, Tuffet S, Lukaszewicz AC, Laplace C, Zucman N, Pocard M, Costaglioli B, Msika S, Duranteau J, Payen D, Dreyfuss D, Hajage D, Ricard JD. Prone positioning in acute respiratory distress syndrome after abdominal surgery: a multicenter retrospective study : SAPRONADONF (Study of Ards and PRONe position After abDOmiNal surgery in France). Ann Intensive Care. 2017 Dec;7(1):21. doi: 10.1186/s13613-017-0235-z. Epub 2017 Feb 24. PMID 28236174
- [Derived] Walter T, Zucman N, Mullaert J, Thiry I, Gernez C, Roux D, Ricard JD. Extended prone positioning duration for COVID-19-related ARDS: benefits and detriments. Crit Care. 2022 Jul 8;26(1):208. doi: 10.1186/s13054-022-04081-2. PMID 35804453